CLINICAL TRIAL: NCT01990261
Title: The Survival of Non-Small Cell Lung Carcinoma EGFR Non-mutated (Wild Type) Patients Treated With Erlotinib (TARceva) After the Failure of at Least One Chemotherapy Regimen
Brief Title: A Study to Assess the Survival of Non-small Cell Lung Cancer Patients Treated With Tarceva After Failed Chemotherapy Treatment
Acronym: STAR
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28496
Record Dates: First submitted 2013-10-31; First posted 2013-11-21 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-06

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Erlotinib: Participants diagnosed with locally advanced or metastatic non-small cell lung with known carcinoma epidermal growth factor receptor (EGFR) status received erlotinib at a dose determined by the investigator, guided by the recommendation in the Summary of Product Characteristics.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib at a dose determined by the investigator, guided by the recommendation in the Summary of Product Characteristics.
  Other Names: Tarceva

SUMMARY:
This study will evaluate the survival of non-small cell lung cancer (wild-type EGFR) participants treated with Tarceva after at least one failed chemotherapy treatment, and the impact of prior chemotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/= 18 years
* Histologically documented locally advanced, metastatic, or recurrent non-small cell lung carcinoma with wild-type EGFR eligible for Tarceva treatment.
* At least one failed chemotherapy treatment.

Exclusion Criteria:

- Unknown EGFR mutation status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with locally advanced, metastatic or recurrent non-small cell lung carcinoma with wild-type EGFR.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 participants were enrolled in 13 centers in Romania.
Period: Overall Study
Arm/Group | Erlotinib
Started | 33
Treated | 29
Completed | 8
Not Completed | 25
Not completed — Death Before Treatment Start | 2
Not completed — Death due to Disease Progression (PD) | 10
Not completed — Death From other Causes | 1
Not completed — Disease Progression (PD) | 8
Not completed — PD Before Treatment Start | 1
Not completed — Dossier not Approved | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
Age, Customized [Number; unit: participants]
  From 18 to 60 years | 10
  60 years and older | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at Month 6
Time Frame: Month 6
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
percentage of participants | 33.3

2. Primary Outcome: Survival Rate at Month 12
Time Frame: Month 12
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
percentage of participants | 15.2

3. Primary Outcome: Progression Free Survival (PFS) at Month 6
Description: PFS is defined as the time from inclusion in the study to the disease progression or death whichever occurs first. Disease progression was determined according to local treatment guidelines.
Time Frame: From inclusion up to disease progression or death whichever occurs first (up to 6 months)
Population: Analysis was performed on all enrolled participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
days | 101.0 [55.194 to 146.806]

4. Primary Outcome: Progression Free Survival (PFS) at Month 12
Description: as for outcome 3
Time Frame: From inclusion up to disease progression or death whichever occurs first (up to 12 months)
Population: Analysis was performed on all enrolled participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
days | 121.0 [62.862 to 179.138]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from first administration of study drug until death from any cause.
Time Frame: Up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Mean (Standard Error); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
days | 74.788 (20.823)

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
percentage of participants | 23

7. Secondary Outcome: Overall Survival According to Prior Chemotherapy Treatment.
Description: Prior chemotherapy treatment is presented as reported by the investigators.
Time Frame: Up to 12 months
Population: Analysis was performed on all enrolled participants.
Measure: Mean (Standard Error); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 33
days
  Carboplatin & Gemcitabine (n=7) | 191.857 (41.756)
  Nabelvina & Carboplatin (n=1) | 80.000 (0.000)
  Carboplatin (n=1) | 138.000 (0.000)
  Carboplatin & Alimta (n=1) | 63.000 (0.000)
  Carboplatin & Vinorelbine (n=1) | 440.000 (0.000)
  Carboplatin & Docetaxel (n=2) | 222.500 (113.500)
  Carboplatin & Paclitaxel (n=4) | 184.875 (81.771)
  Docetaxel, Gemcitabine & Cisplatin (n=1) | 135.000 (0.000)
  Cisplatin & Paclitaxel (n=2) | 268.000 (61.000)
  Docetaxel (n=1) | 115.000 (0.000)
  Gemcitabine (n=1) | 30.000 (0.000)
  Gemzar & Carboplatine (n=3) | 127.667 (39.725)
  Paclitaxel & carboplatin (CBDCA) (n=1) | 80.000 (0.000)
  Taxol & Carboplatin (n=1) | 314.000 (0.000)
  Taxotere (n=1) | 336.000 (0.000)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 3/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=33)
Ischaemic limb pain (Vascular disorders) | 1
Blood bilirubin increased (Investigations) | 1
Sudden death (General disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Disease progression (General disorders) | 3
Ischaemic stroke (Nervous system disorders) | 1
Pleural neoplasms (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=33)
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.